CLINICAL TRIAL: NCT04403568
Title: Phase I Clinical Trial Testing the Synergism of Phytonutrients, Curcumin and Ursolic Acid, to Target Molecular Pathways in the Prostate
Brief Title: Testing the Synergism of Phytonutrients, Curcumin and Ursolic Acid, to Target Molecular Pathways in the Prostate
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No subjects were enrolled in this study, the PI will seek funding and revise the protocol for resubmisson at a later date
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20190735H
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ursolic Acid; Curcumin

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to one of 3 cohorts, starting with cohort 1 and progressing to cohort 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ursolic Acid (Experimental): Administration of Ursolic Acid to subjects who are scheduled to undergo radical prostatectomy
  Interventions: Drug: Ursolic Acid
- Curcumin (Experimental): Administration of Curcumin to subjects who are scheduled to undergo radical prostatectomy
  Interventions: Drug: Curcumin
- Ursolic Acid and Curcumin (Experimental): Administration of Ursolic Acid and Curcumin to subjects who are scheduled to undergo radical prostatectomy
  Interventions: Drug: Ursolic Acid; Drug: Curcumin

INTERVENTIONS:
Drug: Ursolic Acid — Ursolic Acid 150mg
  Arms: Ursolic Acid; Ursolic Acid and Curcumin
Drug: Curcumin — Curcumin 600mg
  Arms: Curcumin; Ursolic Acid and Curcumin

SUMMARY:
A proof of concept clinical trial to assess the synergism of curcumin (CURC) and ursolic acid (UA). Before further testing within formal cancer clinical trials, we must (1) evaluate the bioavailability and safety, (2) confirm the presence of metabolites in the target organ, and (3) validate the appropriate mechanism of effect

DETAILED DESCRIPTION:
Once a subject is identified that may meet eligibility criteria, the physician and/or study investigators will be alerted to the potential candidate and will introduce the study to the patient at their standard of care (SOC) appointment or via telephone. Patients will be given the option for enrollment and if they agree, informed consent will be discussed and obtained provided they meet all inclusion/exclusion criteria. Following informed consent, subjects will be assigned to one of the following cohorts:

Cohort 1:

• Ursolic Acid (150 mg) BID (twice a day)

Cohort 2:

• Curcumin (600 mg) BID

Cohort 3:

• Ursolic Acid (150 mg) and Curcumin (600 mg) BID

The study team aim to enroll 10 subjects who will complete the study into each cohort for a total of 30 completers. Subjects will be enrolled on a rolling basis with the first ten subjects assigned to Cohort 1, the next ten subjects assigned to Cohort 2, and the last 10 subjects assigned to Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

* Have proven diagnosis of prostate cancer with Gleason Group 3 or lower and planning to undergo radical prostatectomy
* Be able to give informed consent
* Be age 18 or older
* Able to stop supplements

Exclusion Criteria:

* Unable to give informed consent
* Age < 18
* High-risk prostate cancer or suspected metastasis
* Unable to swallow pills
* Unable to stop supplements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number, frequency, duration, and relation of toxicity events | Baseline to 8 weeks
  Safety will be compared to evaluate the number, frequency, duration, and relation of toxicity events to CURC/UA combination, as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v 4.03.
Peak serum concentration | Baseline to 8 weeks
  Dose response curve representing the pharmacokinetic parameter peak serum concentration (Cmax) of ursolic acid, curcumin, and their metabolites will be graphed.
Time to reach peak serum concentration | Baseline to 8 weeks
  The pharmacokinetic parameter, the area under the curve (Tmax) representing the time it takes to reach Cmax of ursolic acid, curcumin, and their metabolites will be graphed.
Half-life | Baseline to 8 weeks
  The pharmacokinetic parameter, half-life of ursolic acid, curcumin, and their metabolites will be graphed.

SECONDARY OUTCOMES:
Levels of UA, CURC, and metabolites in prostate tissue | Baseline to 8 weeks
  Identify the presence and levels of UA, CURC and their metabolites in prostate tissue using HPLC.
Immunohistochemistry measurement | Baseline to 8 weeks
  Immunohistochemistry of proportion of nuclear p65 NFkB staining before and after prostatectomy on FFPE samples will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Liss, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data will be available upon completion of the study for approx. 1 year.
Access Criteria: Access granted upon request.